CLINICAL TRIAL: NCT02112851
Title: A Randomized, Placebo-controlled, Double-blind, Crossover Trial to Investigate the Effects of Acute Processed Whole Orange Consumption on Postprandial Glycemic Responses in Healthy Men
Brief Title: Processed Orange and the Glycemic Response
Acronym: POGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1326
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Maximum Observed Plasma Glucose Concentration (Cmax)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Orange flavored beverage (Placebo Comparator): 240ml orange beverage
  Interventions: Other: Orange flavored beverage
- Orange flavored beverage - Test1 (Experimental): 240ml processed whole orange low dose
  Interventions: Other: Orange flavored beverage
- Orange flavored beverage - Test2 (Experimental): 240ml processed whole orange high dose
  Interventions: Other: Orange flavored beverage

INTERVENTIONS:
Other: Orange flavored beverage — Intervention involves consumption of one beverage of 240ml following baseline measurements

SUMMARY:
Randomized, placebo controlled, double blind, postprandial crossover study in male subjects. 3 intervention arms, consisting of a control (Product A), a low dose processed whole orange (Product B) and a high dose processed whole orange (Product C), to determine the effect of the interventions on the primary endpoint of postprandial glycemia. Secondarily, plasma insulin concentrations will be quantified.

DETAILED DESCRIPTION:
The study design is a randomized, placebo controlled, double-blind, crossover. This trial will include 33 subjects randomized to receive products A, B or C [240 mL (255 g)]. Subjects will be randomly assigned to one of 6 sequences of 3 interventions. After the initial screening visit, subjects will visit the Clinical and Translational Research Center (CTRC) the Tufts Translational and Clinical Science Institute (CTSI) on three separate occasions. Following each intervention day there will be a two week wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Males (due to potential hormonal fluctuations in female subjects) aged 30-65 y
* BMI: 25-29.9 kg/m2
* Not diabetic [diagnosed or fasting glucose >7 mmol/L (126 mg/dL)] or suffer from other endocrine disorders
* Not having suffered a myocardial infarction/stroke in the past 12 mo
* Not suffering from renal or bowel disease or have a history of choleostatic liver or pancreatitis
* Not on drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* No history of alcohol misuse
* Not planning or on a weight reducing regime
* Not taking any fish oil, fatty acid or vitamin and mineral supplements
* Non smokers

Exclusion Criteria:

* Females
* Use of medications known to affect lipid metabolism, i.e., hypolipidemic or cholesterol-lowering agents (e.g., Pravastatin, Simuvustatin)
* Use of (>2x/wk) medication for inflammation or hypercoagulation

  * Anticoagulants (Warfarin)
  * Inflammation - NSAID's (Tiaprofenic acid, Sulindac, Ibuprofen), Corticosteroids (Betamethasone)
* Regular use (>2x/wk) of any acid-lowering medications, laxatives or anti-diarrheal medications (prescription or over-the-counter [OTC])
* Use of medications known or suspected to influence blood pressure, including beta-adrenergic blocking agents (oral or ocular) (e.g., Sotalol, Bisoprolol), beta-adrenergic drugs, calcium channel blocking agents (Amlodipine, Nicardipine), angiotensin converting enzyme (ACE) inhibitors (Captopril, Cilazapril), angiotensin receptor blocking agents (Valsartan), nitrates, diuretics (Chlortalidone), venlafaxine and sibutramine, decongestants or chloroquine
* Systolic blood pressure >150 mmHg and/or diastolic blood pressure >95 mmHg
* CVD including coronary artery disease, left ventricular hypertrophy, congestive heart failure, cerebrovascular disease, stroke, peripheral vascular disease or dysautonomia
* Gastrointestinal diseases conditions or medications influencing gastrointestinal absorption including active peptic ulcer disease, treatment with acid-lowering drugs or inflammatory bowel disease
* Renal or chronic kidney disease due to any condition, renovascular disease, history of nephrolithiasis or serum creatinine >1.5 mg/dL
* Endocrine disorders including diabetes [fasting blood glucose >7 mmol/L (126 mg/dL) or current pharmacologic treatment for diabetes], untreated thyroid disease, adrenal disease, pheochromocytoma, parathyroid disease or hyperuricemia
* Rheumatologic diseases including gout or inflammatory arthritis
* Active treatment for cancer of any type (except basal cell carcinoma)<1 y
* Regular use of oral steroids except topical OTC steroids
* Regular use of any dietary supplements containing vitamins, minerals, herbal or other plant-based preparations, fish oil supplements (including cod liver oil) or homeopathic remedies. However, subjects who are willing to refrain from the use of these supplements for 1 mo prior to their initial visit (Visit 3) may be considered eligible.
* Usual daily ethanol intake of>2 drinks (24 oz beer, 8 oz wine, 2 oz hard liquor)
* Cigarette smoking and/or nicotine replacement use. However, subjects who have stopped using these products for 1 y prior to their initial visit (Visit 1) may be considered eligible.
* Illicit drug use
* Infrequent (<3/wk) or excessive (>3/d) number of regular bowel movements
* Specific laboratory blood or urine analysis parameters of:

  * Creatinine > 1.5 mg/dL
  * Electrolytes, calcium, phosphorous - out of normal ranges
  * ALT and AST >1.5 nmol
  * Total bilirubin - above normal range
  * Triglycerides ≥300 mg/dL
  * Fasting glucose ≥126 mg/dL
  * CBC: HCT outside of normal NEL reference ranges at the discretion of the study physician
  * WBC, PLT - outside of normal NEL reference ranges Strict vegetarians
* Those on or planning a weight reducing regime
* Unable to consume study meals or products
* Subjects with larger than 5 kg weight loss in the last 3 months.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma glucose concentration (Cmax) | 0-8 hours

SECONDARY OUTCOMES:
Maximum observed plasma insulin concentration (Cmax) | 0-8 hours
Area under the curve (AUC) of glucose and insulin and the time to reach Cmax gluc (Tmax gluc) and Cmax ins (Tmax ins) | 0-8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States